CLINICAL TRIAL: NCT00760669
Title: Post Marketing Surveillance of Remicade in Ankylosing Spondylitis, Rheumatoid Arthritis, Psoriatic Arthritis and Psoriasis Patients
Brief Title: An Observational Study of Infliximab Injection in Ankylosing Spondylitis, Rheumatoid Arthritis, Psoriatic Arthritis and Psoriasis Participants
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100768; REMICADEAKS4004 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Spondylitis, Ankylosing; Arthritis, Rheumatoid; Psoriasis; Arthritis, Psoriatic
Keywords: Spondylitis, Ankylosing; Arthritis, Rheumatoid; Psoriasis; Arthritis, Psoriatic; Infliximab; Remicade
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Rheumatoid; Psoriasis; Arthritis, Psoriatic | interventions — Infliximab; Observation; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Receiving Infiximab: Participants with rheumatoid arthritis (RA), ankylosing spondylitis (AS) and psoriatic arthritis (PA) receiving infliximab injection will be observed.
  Interventions: Drug: Infliximab; observational study; Drug: Methotrexate; observational study

INTERVENTIONS:
Drug: Infliximab; observational study — This is an observational study. Participants with RA, AS and PA receiving induction intravenous infusions (a fluid or a medicine delivered into a vein by way of a needle) of infliximab will be observed. Participants with RA will receive infliximab 3 milligram per kilogram (mg/kg) as an intravenous infusion over a 2-hour period followed by additional 3 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks (maintenance) thereafter up to 30 weeks. Participants with AS and PA will receive 5 mg/kg infliximab as an intravenous infusion over 2-hour period followed by additional doses at 2 and 6 weeks up to 24-30 weeks and 30 weeks, respectively.
  Other Names: Remicade Injection
Drug: Methotrexate; observational study — Participants with RA will receive methotrexate based on physician's clinical judgement.

SUMMARY:
The purpose of this observational study is to evaluate the safety and effectiveness of infliximab injection under actual conditions of use in participants, and to learn more about its adverse events.

DETAILED DESCRIPTION:
This is an observational, prospective (study following participants forward in time) study to assess safety and efficacy of infliximab injection under post-marketing use and identify problems related to adverse events in participants with ankylosing spondylitis (chronic inflammatory condition affecting the axial joints), rheumatoid arthritis (chronic systemic disease, primarily of the joints, marked by inflammatory changes in the synovial membranes and articular structures), psoriasis (scaly skin rash) and psoriatic arthritis (a type of inflammatory arthritis associated with psoriasis). Participants with rheumatoid arthritis will receive 6 doses of infliximab 3 milligram per kilogram (mg/kg) as an intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) at Week 0, 2, 6 and will be observed for 30 weeks; and those with ankylosing spondylitis, psoriasis and psoriatic arthritis will also receive 6 doses of injection and will be observed for 24 to 30 weeks. Efficacy will be evaluated by Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Erythrocyte Sedimentation Rate (ESR), C-reactive protein (CRP), Psoriasis Area and Severity Index (PASI), swollen joint counts and tender joint count. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with ankylosing spondylitis who did not show adequate response to general treatments and with increased serological indices related to severe axial symptoms and inflammation
* Participants with rheumatoid arthritis who show insufficient response to disease modifying antirheumatic drug (DMARD) including methotrexate
* Participants with serious, active and progressive disease not previously treated with methotrexate or other DMARD
* Participant with moderate to serious plaque psoriasis who are unresponsive, contra indicant or intolerable to the systemic therapy including cyclosporine, methotrexate or Psoralen Ultra-Violet A (PUVA)
* Participant with active, progressive, psoriatic arthritis who have shown insufficient response to DMARD treatment

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participant with ankylosing spondylitis, rheumatoid arthritis, psoriasis and psoriatic arthritis will be observed at rheumatology departments in university or general hospitals where they are commonly treated.
Sampling Method: Non-Probability Sample
Enrollment: 1061 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Receiving Infliximab: Participants with rheumatoid arthritis (RA), ankylosing spondylitis (AS) and psoriatic arthritis (PA) receiving induction intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) of infliximab at Week 0, 2, and 6 were observed. Dosage and infusion intervals of infliximab were employed in accordance to the summary of product characteristics: participants with RA received infliximab 3 milligram per kilogram (mg/kg) as an intravenous infusion over a 2-hour period followed by additional 3 mg/kg infusion doses at 2 and 6 weeks after the first infusion, then every 8 weeks (maintenance) thereafter up to 30 weeks along with methotrexate, participants with AS and PA received 5 mg/kg infliximab as an intravenous infusion over 2-hour period followed by additional doses at 2 and 6 weeks up to 24-30 weeks and 30 weeks, respectively.
Period: Overall Study
Arm/Group | Participants Receiving Infliximab
Started | 1061
Completed | 1031
Not Completed | 30
Not completed — Not assessed for overall improvement | 18
Not completed — Participants missing efficacy assessment | 6
Not completed — Participants with overlapping cases | 1
Not completed — Took drug before entering in contract | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were performed on safety analysis set. Data presented only for 1055 participants as they were part of safety analysis set. Safety analysis set included all participants who received at least 1 dose of study medication.
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 1055
Age Continuous [Mean (Standard Deviation); unit: years] | 39.32 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 363
  Male | 692

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 30
Description: The BASDAI is a validated self-assessment tool used to assess disease activity in participants with ankylosing spondylitis. It consists of 6 items measuring fatigue, spinal pain, joint pain, areas of localized tenderness, intensity of morning stiffness and duration of morning stiffness. First 5 items are scored on a 10 millimeter (mm) Visual Analog Scale (VAS) ranging from 0 mm=none to 10 mm=severe; and sixth item is scored on VAS ranging from 0=0 hours to 10=2 or more hours. The total BASDAI score ranges from 0 (none) to 10 (very severe).To give each symptom equal weighting, the average of the 2 scores relating to morning stiffness was taken. The resulting 0 to 50 score is divided by 5 to give a final BASDAI score. BASDAI total score = 0.2 (Item 1 + Item 2 + Item 3 + Item 4 + Item 5/2 + Item 6/2).
Time Frame: Baseline and Week 30
Population: The efficacy assessment analysis set included all participants who were assessed for efficacy assessment. Here 'N' (number of participants analyzed) signifies participants who were diagnosed with ankylosing spondylitis and were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 705
Millimeter
  Baseline | 7.52 (6.68)
  Change at Week 30 | -5.23 (4.51)

2. Primary Outcome: Change From Baseline in Erythrocytic Sedimentation Rate (ESR) at Week 30
Description: The ESR is a laboratory test that provides a non-specific measure of inflammation. It assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm per hour. A higher rate indicated inflammation.
Time Frame: Baseline and Week 30
Population: The efficacy assessment analysis set included all participants who were assessed for efficacy assessment. Here 'N' (number of participants analyzed) signifies participants who were diagnosed with rheumatoid arthritis or psoriatic arthritis and were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimeter per hour
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 248
Millimeter per hour
  Baseline | 60.75 (29.84)
  Change at Week 30 | -21.80 (29.88)

3. Primary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 30
Description: The CRP is acute serum protein released from liver. It is associated with low hemoglobin or erythropoetic resistance. The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is less than 1 milligram per deciliter (mg/dl). A decrease in the level of CRP indicated reduction in inflammation and therefore improvement.
Time Frame: Baseline and Week 30
Population: The efficacy assessment analysis set included all participants who were assessed for efficacy assessment. Here 'N' (number of participants analyzed) signifies the participants who were diagnosed with rheumatoid arthritis or psoriatic arthritis and were evaluated for this measure.
Measure: Mean (Standard Deviation); unit: Milligram per deciliter
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 262
Milligram per deciliter
  Baseline | 7.94 (14.04)
  Change at Week 30 | -4.81 (11.23)

4. Primary Outcome: Change From Baseline in Number of Swollen Joints at Week 30
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit and scored on a scale ranging from 0 to 2, where 0=no swelling, 1=swelling, but bony landmarks seen and 2=swelling but bone marks not seen.
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 239
Swollen joints
  Baseline | 9.75 (6.53)
  Change at Week 30 | -5.46 (6.02)

5. Primary Outcome: Change From Baseline in Number of Tender Joints at Week 30
Description: Number of tender joints was determined by examination of 28 joints and identifying when tenderness was present. The number of tender joints was recorded on the joint assessment form at each visit and scored on a scale ranging from 0 to 3, where 0=no pain, 1=mild, 2= moderate and 3=severe.
Time Frame: Baseline and Week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 240
Tender joints
  Baseline | 13.31 (7.75)
  Change at Week 30 | -7.35 (7.42)

6. Primary Outcome: Change From Baseline in Participants With Psoriasis Area and Severity Index (PASI) at Week 30
Description: The PASI is combined assessment of lesion severity and area affected into single score; range: 0=no disease to 72=maximal disease. Body is divided into 4 sections (head, arms, trunk and legs); each area is scored by itself and scores were combined for final PASI. For each section percent area of skin involved was estimated: 0 (0%) to 6 (90 - 100%), and severity was estimated by clinical signs: erythema, thickness, and scaling; scale: 0 (none) to 4 (severe). Final PASI=sum of severity parameters for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
Time Frame: Baseline and Week 30
Population: Data was not evaluated as only 1 participant with psoriatic arthritis was enrolled in this surveillance and no PASI evaluation was done for it.
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 0

7. Primary Outcome: Overall Efficacy Assessment
Description: The level of improvement in symptom before and after the administration of the drug was assessed as per Investigator's discretion and the overall efficacy was assessed based on this result. The level of improvement in disease was assessed in three steps: improved, unchanged and aggravated as per Investigator's discretion.
Time Frame: Baseline up to Week 30
Population: The efficacy assessment analysis set included all participants who were assessed for efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 1031
Participants
  Improved | 948
  Unchanged | 59
  Aggravated | 24

8. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Week 30
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 1055
Participants
  AEs | 106 (7.75)
  SAEs | 12 (7.42)

9. Primary Outcome: Number of Participants With Unexpected Adverse Events
Description: Unexpected adverse events include those not listed in the approved product information and not described as precautions or warnings.
Time Frame: Baseline up to Week 30
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 1055
Participants | 28 (7.42)

10. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events for which the Investigator had not described the causal relationship to trial medication as "not related".
Time Frame: Baseline up to Week 30
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 1055
Participants | 59 (7.75)

11. Primary Outcome: Number of Participants With Adverse Events (AEs) Caused by Drug Misuse, Abuse and Drug Interaction
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Drug abuse is defined as the use of the study drug for a non-therapeutic effect, misuse was defined as use of the study medication in a way that was not prescribed and drug interaction was defined as a chemical or physiological reaction that can occur when 2 different drugs are taken together.
Time Frame: Baseline up to Week 30
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Participants Receiving Infliximab
Number analyzed (Participants) | 1055
Participants | 48

ADVERSE EVENTS:
Time Frame: Baseline up to 30 weeks
Arm/Group | Participants Receiving Infliximab
Serious Adverse Events (participants affected / at risk) | 12/1055
Other Adverse Events (participants affected / at risk) | 95/1055
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Infliximab (N=1055)
Cellulitis (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Disseminated tuberculosis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Spinal shock (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Glaucoma (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Receiving Infliximab (N=1055)
Nasopharyngitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 6
Folliculitis (Infections and infestations) | 2
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic tonsillitis (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pelvic abscess (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Epigastric discomfort (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Hepatic enzyme increased (Investigations) | 12
Blood pressure increased (Investigations) | 1
Hepatic enzyme abnormal (Investigations) | 1
LE cells present (Investigations) | 1
Chills (General disorders) | 4
Chest discomfort (General disorders) | 3
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 3
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Hepatitis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Palpitations (Cardiac disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Pregnancy of partner (Social circumstances) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) cannot provide any trial related information to external parties' without mutual agreement with the Sponsor. This is valid even after the contract is canceled.